CLINICAL TRIAL: NCT03967353
Title: Study on the Management Model of "Home Treatment" for Tuberculosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, FengLing Mi, vice director of office of academic research, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D 181100000418002
Record Dates: First submitted 2019-05-23; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Tuberculosis; Home Treatment Management; Infection Control
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Treatment Group (No Intervention): Routine treatment group(6 months treatment regimen-2HRZE/4HR); Routine health education; Dose-taken supervised by family members
- Intervention Group (Experimental): Using mobile technology management means to manage newly treated smear-positive tuberculosis patients, to guide patients'treatment, infection control, doctor-patient communication, and to strengthen health education on infection control of patients.
  Interventions: Behavioral: New management mode intervention

INTERVENTIONS:
Behavioral: New management mode intervention — Patients in routine treatment group use "TB assistant APP". Medical staff strengthen health promotion of the patients,including, infection control, doctor-patient communication, etc.
  Arms: Intervention Group

SUMMARY:
This project aims to standardize the management of "home treatment" for tuberculosis patients, improve the compliance of patients with treatment, reduce the risk of transmission, and study the establishment of "home treatment" management model for tuberculosis patients.

DETAILED DESCRIPTION:
The project intends to optimize the standardized management framework and process of "home treatment" for tuberculosis patients by introducing mobile Internet technology as a means of patient management and formulating "home treatment" infection control norms, and ultimately form a management model suitable for "home treatment" for tuberculosis patients.Through prospective study to evaluate the effect of this model on the treatment compliance of "home treatment" patients and the impact on tuberculosis infection and incidence of close contacts, so as to further improve the "home treatment" management model. The research results of this project will provide policy basis for Beijing to formulate "home treatment" management of tuberculosis progress.

ELIGIBILITY:
Inclusion Criteria:

Pathogenic Comfirmed Positive TB patients New Pathogenic Positive Pulmonary Tuberculosis Patients Treated by Home Treatment TB assistant APP user

Exclusion Criteria:

Unconscious Unable to answer questions

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2018-03-22 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
treatment adherence | 6 months for each patient
  to compare the adherence rate of the two groups

SECONDARY OUTCOMES:
treatment success rate | 6 months for each patient
  to compare the success rate of the two groups

CONTACTS AND LOCATIONS:
Overall Officials: fengling Mi, Master, Study Director — Beijing Chest Hospital, Capital Medical University
Locations (1):
- Beijing Chest Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
To share the data to main researchers.